CLINICAL TRIAL: NCT05269277
Title: Health System Methods to Improve Nursing Retention Amidst Ongoing COVID-19 Pandemic: a Mixed Method Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Poudre Valley Health System (Other)
Responsible Party: Principal Investigator, Claire Aksamit, Investigator, Poudre Valley Health System
Other Study IDs: 21-4768
Record Dates: First submitted 2022-03-01; First posted 2022-03-07 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Motivational Factors for Nurse Retention; Nurse Well-being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a mixed-method exploratory study with the aim to determine an objective compensation or mechanism of support from a healthcare system standpoint to aid in retention of nursing staff amidst the ongoing COVID-19 pandemic. It will include semi-structured qualitative interviews of current and prior nursing staff from the Trauma/Surgical floor, Progressive Care Unit, and ICU, in addition to Trauma/Surgical unit and system administrators; the second portion of the study will include a quantitative survey distributed via email to current nurses on the Trauma/Surgical floor, Progressive Care Unit, and ICU to assess ranked priority of additional mechanisms of support to improve intention of retention.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses on the Trauma/Surgical floor, Surgical Progressive Care Unit, or Surgical ICU who are currently working or who have worked bedside in the past 24 months
* Adult hospital administrative staff

Exclusion Criteria:

* Non-Registered nurses (ie. CNAs, LPNs)
* RNs without clinical bedside experience in the past 24 months
* RNs working on other units beside the Trauma/Surgical floor, Surgical Progressive Care Unit, or Surgical ICU

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants for the qualitative interviews will include current bedside nursing and clinical administrative staff at UCHealth - Medical Center of the Rockies on the Trauma/Surgical floor, the Surgical Progressive Care Unit, and the Surgical ICU. Other participants will also include prior nurses who have left their job on these respective units in the prior 24 months. Registered nurses, men and women, day-time and night-time nurses, full-time versus part-time nurses, and those with variable lengths of experience will be incorporated who have been or are currently involved with direct patient care during the COVID-19 pandemic. The quantitative survey will be distributed to all current nurses on the above listed units.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify a common mechanism or implementation to improve intention of retention or nurses amongst the Trauma/Surgical units amidst COVID-19 | 24 months
  The goal is to identify a common theme amongst nurses on the Trauma/Surgical units regarding a means of compensation or action item from the healthcare system to improve intention of retention amidst ongoing COVID-19 pandemic. Obtaining this is two-fold, to include qualitative interviewing with nurses on the affected units first-hand with subsequent transcription and coding to identify common themes; and a widely distributed quantitative survey to assess ranked priorities to implement to improve intention of retention.

SECONDARY OUTCOMES:
Commonly-identified challenges nurses are facing on a Trauma/Surgical unit during COVID-19 | 24 months
  The goal is to identify common challenges nurses on Trauma/Surgical units during COVID-19. This will primarily be obtained via qualitative interviewing of nurses on the affected unit first-hand to discuss the most challenging parts of their jobs, in particularly during COVID-19, subsequently followed by transcription and coding and analysis to identify common themes.
Commonly-identified support mechanisms implemented by the healthcare system that have aided in intention of retention of nurses on a Trauma/Surgical unit during COVID-19 | 24 months
  The goal is to identify common interventions the healthcare systems has provided that has helped with intention of retention of nursing staff during COVID-19. To obtain this, qualitative interviewing will be done speaking to affected nurses first-hand, following by subsequent transcription and coding and data analysis to identify these common themes.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Aksamit, Principal Investigator — University of Colorado Health
Locations (1):
- UCHealth - Medical Center of the Rockies, Loveland, Colorado, United States

DOCUMENTS (2):
  • Study Protocol (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT05269277/Prot_000.pdf
  • Informed Consent Form (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT05269277/ICF_001.pdf